CLINICAL TRIAL: NCT01628445
Title: Phase 3 Study of Liraglutide in Individuals With Type 2 Diabetes Using Insulin
Brief Title: Study of Liraglutide in Individuals With Type 2 Diabetes Using Insulin
Acronym: SAIL
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Error made by local pharmacy caused mixed randomization of 20 participants
Sponsor: University of Manitoba (Other)
Collaborators: Novo Nordisk A/S (Industry)
Responsible Party: Principal Investigator, Dr. Vincent Woo, Assistant Professor, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: U1111-1126-3937
Record Dates: First submitted 2012-06-21; First posted 2012-06-26 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Type 2 Diabetes
Keywords: Diabetes; Insulin
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Liraglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- liraglutide (Active Comparator): liraglutide 1.8 mg injected once daily
  Interventions: Drug: liraglutide
- Placebo injection (Placebo Comparator)
  Interventions: Drug: placebo injection

INTERVENTIONS:
Drug: liraglutide — liraglutide titrated to 1.8 mg sc daily
  Other Names: Victoza
  Arms: liraglutide
Drug: placebo injection — placebo injected sc daily volume equal to active comparator
  Other Names: Placebo
  Arms: Placebo injection

SUMMARY:
Liraglutide is a GLP1 agonist used in the treatment of Type 2 diabetes and is is asociated with improved blood glucose control, weight loss and low rates of hypoglycemia when used alone or in combination with metformin. Liraglutide has not been extensively tested in people with type 2 diabetes who are taking relatively large doses of insulin (>50 U/day). Often these patients are insulin resistant and despite using large doses of insulin are not able to achieve glucose targets. The rationale for this study is to assess if the addition of liraglutide in addition to usual care versus placebo can improve blood glucose levels in people not achieving a target HbA1C of less than 7.0%.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* BMI≤45 kg/m2
* A1c ≥7.5% and ≤10.5%

Exclusion Criteria:

* type 1 diabetes
* symptoms of poorly controlled diabetes
* eGFR <50 ml/min/1.73m2

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2012-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change in A1c | Baseline to 24 wks

SECONDARY OUTCOMES:
Percentage of patients experiencing hypoglycemia | Baseline and 24 weeks
Change in Systolic Blood pressure | Baseline and 24 weeks
Change in diastolic blood pressure | Baseline and 24 weeks
Change in waist circumference | Baseline and 24 weeks
Change in body weight | Baseline and 24 weeks
Change in heart rate | Baseline and 24 weeks
Change in lipid profile | Baseline and 24 weeks
Diabetes Treatment Satisfaction | Baseline, 12 weeks and 24 weeks
Percentage of patients achieving A1C < or equal to 7% | Baseline and 24 weeks
Change in fasting blood glucose | Baseline adn 24 weeks
Occurence of undetected hypoglycemia as measured by continuous glucose monitoring | Baseline, 12 weeks and 24 weeks
Postprandial glucose reduction through measurement of 7 point glucose profile | Baseline, 4 weeks, 12 weeks and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vincent C Woo, MD FRCPC, Principal Investigator — University of Mantioba
Locations (1):
- Winnipeg Regional Health Authority Health Sciences Centre Winnipeg Diabetes Research Group, Winnipeg, Manitoba, Canada